CLINICAL TRIAL: NCT02310945
Title: Pain Sensitization and the Risk of Poor Outcome Following Physiotherapy for Knee Osteoarthritis: A Protocol for a Prospective Cohort Study
Brief Title: Pain Sensitization and Outcome Following Physiotherapy in Patients With Knee Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Sponsor
Other Study IDs: HPF/2013/44
Record Dates: First submitted 2014-11-28; First posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Knee Osteoarthritis
Keywords: pain; central nervous system sensitization; physiotherapy
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Knee osteoarthritis: People with moderate/severe symptomatic knee osteoarthritis referred for physiotherapy
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Individualised programme for each patient in line with current clinical guidelines. May include education, exercise (strengthening, range of motion exercise, aerobic), lifestyle advice and manual therapy

SUMMARY:
Pain is the dominant symptom of knee osteoarthritis and recent evidence suggests factors outside of local joint pathology, such as pain sensitization, can contribute significantly to the pain experience. It is unknown how pain sensitization influences outcomes from commonly employed interventions such as physiotherapy.

The aims of this study are, firstly to identify people with knee OA who display signs and symptoms associated with pain sensitization using clinical tools and quantitative sensory testing. Secondly, we will investigate if indications of pain sensitization at baseline are associated with poor outcome following physiotherapy.

Methods and analysis:

This is a multi-centre prospective cohort study with 140 participants. Eligible patients with moderate/severe symptomatic knee osteoarthritis will be identified at hospital outpatient clinics. A baseline assessment will provide a comprehensive description of the somatosensory characteristics of each participant by means of clinical examination, quantitative sensory testing and validated questionnaires measuring pain and functional capacity. Participants will then undergo physiotherapy treatment, in line with current clinical guidelines. Follow-up post physiotherapy treatment (estimated to be at 3 months) will assess pain, disability (sub-scales of Western Ontario and McMasters University Score Osteoarthritis Index) and participants' global rating of change. These primary outcome measures will dichotomise participants into treatment 'responders' and 'non-responders' according to the Osteoarthritis Research Society International (OARSI) treatment responder criteria.

For data analysis results from pressure pain thresholds, temporal summation and conditioned pain modulation will create a composite score of pain sensitization. Logistic regression will explore the relationship between response to physiotherapy and pain sensitization at baseline while accounting for various cofounders.

DETAILED DESCRIPTION:
BACKGROUND

The pathophysiology of knee OA pain is complex. Altered processing of nociceptive inputs at spinal and higher brain centers may help explain discrepancies between pain severity and pathological abnormalities in OA. Central sensitization is described as an increased responsiveness of nociceptive neurons at spinal and supraspinal levels to normal or sub-threshold afferent input leading to hyperalgesia. It may also include dysfunction of endogenous pain control systems. Furthermore, peripheral pro-inflammatory mediators and neuropeptides in knee OA can sensitize nociceptors, lowering their threshold for activation. This increased responsiveness of peripheral nociceptors is referred to as peripheral sensitization.

Both peripheral and central nervous system sensitization, clinically referred to as pain sensitization can result can be an enhanced, persistent and more widespread pain response. Recent studies have found the presence of increased pain sensitivity at remote sites, enhanced temporal summation and hypersensitivity to various stimuli to be associated with reports of more severe knee pain symptoms. These studies are cross-sectional and although they link signs of sensitization with greater levels of pain and disability they cannot infer causality.

There is some evidence to suggest increased pain sensitivity negatively affects treatment outcomes. In painful musculoskeletal conditions such as shoulder impingement and lateral epicondylalgia widespread pressure pain sensitivity and thermal hyperalgesia, have been linked with a poorer prognosis. Surgical outcomes for knee osteoarthritis may also be affected with the presence of increased pain sensitivity prior to total knee replacement associated with more persistent pain after surgery.

Physiotherapy is a widely recommended conservative management approach. Studies of prognosis in knee OA have focused on demographic and psychological variable, few studies have focused on factors relating to abnormal pain processing. No longitudinal studies have explored prognostic factors relating to pain sensitization and outcome following physiotherapy. In whiplash associated disorders the presence of sensory hypersensitivity and cold hyperalgesia has been shown to reduce the likelihood of a positive response to physiotherapy treatment. Thus it is conceivable, but currently unproven, that knee OA patients with evidence of pain sensitization have poorer outcomes following physiotherapy.

One obstacle to investigating the implications of pain sensitization is reliably identifying it in the clinical setting. Clinical criteria proposed for assessing central sensitization rely principally on the clinician's subjective interpretation of patient symptoms. Although useful clinically, for research purposes more objective measures are preferable. Due to the complexity of the pain experience it is inadvisable to rely on any single test to reflect peripheral and central pain mechanisms. A multi-tissue assessment using a multi-modal stimuli approach has been advocated, and will be adopted in this study. Recognised features of central and peripheral sensitization previously identified in knee OA patients will be incorporated into this study and these include extended areas of hyperalgesia, enhanced temporal summation, and dysfunctional conditioned pain modulation.

This study will explore clinical outcomes of knee OA (pain, function, patient's global assessment) following physiotherapy, investigating the association between key features of pain sensitization and the likelihood of a poor outcome. Distinguishing patients at risk of a poor outcome can help determine appropriate management strategies in a timely manner.

STUDY AIMS:

The main aims of the study are; firstly to provide a comprehensive description of the somatosensory characteristics of people with pain associated with knee OA (by means of clinical examination, QST, and validated questionnaires measuring pain, functional capacity and quality of life) and secondly, to investigate if the presence of pain sensitization at baseline is associated with poorer response to physiotherapy treatment.

METHODS AND ANALYSIS:

Study design:

A multi-centre observational cohort study with assessments at baseline, at 3 months (on completion of physiotherapy treatment) and at six months will be conducted. Following the baseline assessment for features of pain sensitization all participants will receive usual physiotherapy care. The relationship between pain sensitization and outcomes in terms of pain and disability will be explored through regression analysis.

Setting:

The study will be set in the physiotherapy outpatient departments of three large publicly funded teaching hospitals in Dublin, Ireland.

Participants:

Patients with symptomatic knee OA referred for physiotherapy treatment by a hospital consultant or clinical specialist physiotherapist will be eligible for inclusion.

Healthy controls:

Forty age and gender matched pain-free controls will be recruited. The controls will provide reference data for QST results.

Recruitment procedure:

A consecutive sample of knee osteoarthritis patients with moderate/severe knee pain will be recruited. Potentially eligible participants will be identified at musculoskeletal assessment clinics and from physiotherapy outpatient waiting lists. A feasible recruitment rate is estimated at 12 patients per month with recruitment continuing until the specified numbers are achieved. Those who agree to participate will attend for a baseline assessment prior to commencing physiotherapy treatment. Written informed consent will be obtained before enrolment in the study.

Physiotherapy management:

Physiotherapy treatment will be in line with current clinical guidelines for the management of knee OA. (McAlindon et al., 2014). A workshop led by the principal investigator will be held at each recruitment site prior to study commencement where physiotherapists will receive an update on clinical guidelines and current best evidence on management of knee OA. This will standardise treatment to some degree, but intervention will be individualised at the discretion of the treating physiotherapist.

Assessment

Baseline assessment:

Each baseline assessment will take approximately 50 minutes to complete at the physiotherapy clinic by the principal investigator. Some questionnaires will be posted and completed in advance by participants.

Follow up assessment:

The primary endpoint will be on completion of physiotherapy treatment (this is expected to be at 3 months; estimated duration of a course of physiotherapy treatment).

Six months after enrolment into the study participants will complete a postal questionnaire assessing pain and function. They will exit the study at this point.

Testing procedure:

In order to improve reliability of the assessment and minimise bias standardised assessment procedures will be followed. Studies support the reliability of QST measures where protocols are standardised and both the tester and participant are carefully instructed.

Outcome Variables:

Primary and secondary outcomes are outlined in section below.

Identifying and Quantifying Pain Sensitization:

Abnormal pain pressure thresholds and temporal summation have been previously used for identifying sub-groups of patients with widespread pain hypersensitivity. Conditioned pain modulation (CPM) is reflective of the endogenous inhibitory capacity of the nociceptive system and dysfunction of CPM is associated with syndromes such as fibromyalgia and temporomandibular joint disorder where central sensitization is a recognised hallmark. Pain sensitization will therefore be operationalized by the presence of decreased PPTs and enhanced temporal summation at local (knee) and remote (arm) sites in addition to dysfunctional CPM. The cut-off point for what is abnormal or sensitized will be determined when control data has been gathered and the spread or variability of 'normal' results is seen. Points will be summed to produce a pain sensitization score where a higher score will represent greater pain sensitization.

DATA ANALYSIS PLAN

Data will be analysed using SPSS v 20 (SPSS Inc., Chicago, IL). Descriptive statistics will be calculated for all outcome measures at baseline.

Initial analyses will be exploratory to compare symptom profiles between people who respond to treatment and treatment non-responders. Treatment responders will be categorised by the OMERACT-OARSI responder criteria. Categorical variables will be analysed using chi-square tests. Multivariate analysis of variance (MANOVA) will be used to compare continuous normally distributed variables between responders and non-responders. The Kruskal-Wallis test will be used for comparison of variables that are not normally distributed. A p value of less than 0.05 will be considered significant.

A logistic regression model will be developed to predict response to physiotherapy treatment with 'treatment responder' as the dependant variable. The model will be adjusted for predetermined variables based on the previous literature (age, gender, obesity, socioeconomic status, depressive symptoms, treatment adherence, comorbidities and presence of widespread pain). The pain sensitization score will be entered into the regression model as an independent variable.

Sample size:

The sample size was calculated based on the number of explanatory variables planned for inclusion in the logistic regression model. It is intended to include 8 explanatory variables and allow 15 participants for each explanatory variable. Recruiting 140 participants while allowing for a 20% loss to follow-up should ensure adequate numbers.

Dropouts:

All participants will be followed up on discharge from physiotherapy. Patients will be considered lost to follow-up if they do not complete the primary outcome measure post treatment.

DISCUSSION

To our knowledge this is the first study to examine the effects of pain sensitization on clinical outcomes in response to physiotherapy in patients with knee OA.

There is a lack of a standardized protocol for assessing pain sensitization in the clinical setting. This study selects tests based on their utility in the clinical setting. The results may identify a small selection of outcome measures that are practical for assessing pain sensitization and associated with an increased risk of poor outcome.

This clinically based observational study does not aim to investigate the effects of specific physiotherapy treatments. It will observe people undergoing usual physiotherapy and variation in the intervention is to be expected. Nonetheless an attempt to standardise care to some degree will be made by using current evidence based guidelines and keeping a record of the physiotherapy intervention and adherence for each participant.

Recruiting the participant sample from the secondary care setting will limit the generalizability of study findings to patient populations in primary care.

Given its relatively short follow-up period we cannot infer causality directly from our data with regard to pain sensitization and physiotherapy outcomes. Nonetheless it may point to a relationship worthy of further investigation in order to better understand pain mechanisms in knee OA and optimise physiotherapy outcomes in the future.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis diagnosed by American College of Rheumatology clinical criteria
* Knee pain must be the primary musculoskeletal complaint participant is seeking treatment for
* Pain duration greater than 3 months
* Pain severity ≥ 5/10 on Numerical Rating Scale
* Willing to abstain from simple analgesics and NSAIDs for 24 hours prior to testing
* Willing and able to give full consent

Exclusion Criteria:

* Lumbar or cervical radiculopathy,
* Systematic inflammatory disease,
* Positive screen for diabetic neuropathy
* Past medical history
* Previous surgery or disease of the peripheral or central nervous system,
* Sensory loss secondary to chemotherapy or radiotherapy
* Fibromyalgia
* Chronic fatigue syndrome
* Cognitive or psychiatric disorder interfering with ability to cooperate with assessment
* Injection or physiotherapy treatment for knee joint within previous 3 months
* Taking anti-depressant or anti-convulsant medication

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will be recruited from patients with moderate/severe symptomatic knee OA attending outpatient orthopaedic and rheumatology clinics and referred for physiotherapy treatment by a hospital consultant or clinical specialist physiotherapist.
  At the time of recruitment knee pain must be the participant's primary musculoskeletal complaint they are seeking treatment for, and physiotherapy must be the main treatment being undertaken over the study period
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-10 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Change in response to physiotherapy as measured by the pain and function sub-scales of Western Ontario and McMasters University Score Osteoarthritis Index (WOMAC) and patient's global rating of change. | Baseline & at 3 months (estimated time point for physiotherapy treatment completion)
  These 3 outcome measures will gather data that will be applied to a set of treatment responder criteria by the Outcome Measures in Rheumatology - Osteoarthritis Research Society International (OMERACT-OARSI) to determine a positive response to physiotherapy or a 'treatment responder'

SECONDARY OUTCOMES:
Quantitative sensory testing (pressure pain thresholds, temporal summation, conditioned pain modulation, mechanical detection thresholds) | Baseline
  To describe the somatosensory characteristics of the sample and detect features of pain sensitization
Central Sensitization Inventory | Baseline
  Questionnaire to assess for symptoms not related to the musculoskeletal system but common to central sensitization syndromes
Modified PainDETECT | Baseline
  Questionnaire that records any neuropathic component to patient's symptoms
Centre for Epidemiologic Studies Depression Scale (CES-D) | Baseline
  A measure of depressive symptoms
Overweight/Obesity | Baseline
  Measured by recording participants' waist circumference to height ratio
Manual tender point count | Baseline
  Manual tender point examination to identify tender points according to the American College of Rheumatology criteria for fibromyalgia
EQ-5D 5L | Baseline
  Questionnaire to measure health related quality of life
Self Administered Comorbidity Questionnaire | Baseline
  Questionnaire to record presence of comorbid conditions
Widespread pain | Baseline
  Widespread pain is defined according to the American College of Rheumatology classification criteria using pain drawings marked by participants on a body manikin
Patient adherence monitored over the course of physiotherapy treatment (Sports Injury Rehabilitation Adherence Scale (SIRAS) and Home Exercise Compliance Assessment (HECA) ) | Recorded at each physiotherapy appointment (approx 6 times between 0 and 3 months)
  SIRAS records physiotherapist's perceptions of patient's rehab adherence. HECA is a self-report method for patients to measure their own adherence
Change in medication use and use of co-interventions | At 3 months (estimated time point for physiotherapy treatment completion)
  Any self reported change in medications and co-interventions. Recorded at 3 months using follow-up questionnaire.
Change in knee pain and disability at 6 months | Baseline and at 6 months
  Measured with pain and disability sub-scales of Western Ontario and McMasters University Score Osteoarthritis Index (WOMAC)

CONTACTS AND LOCATIONS:
Overall Officials: Helen O'Leary, BSc Physio, Principal Investigator — University College Dublin; Catherine Doody, BSc Physio, Study Director — University College Dublin; Keith Smart, BSc Physio, Study Chair — St Vincent's University Hospital, Ireland; Niamh Moloney, BSc Physio, Study Chair — University College Dublin
Locations (3):
- Ireland (3):
  - St. James's Hospital, Dublin, Dublin
  - St. Vincent's University Hospital, Dublin, Dublin
  - Tallaght Hospital, Dublin, Dublin

REFERENCES:
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159
- [Background] Finan PH, Buenaver LF, Bounds SC, Hussain S, Park RJ, Haque UJ, Campbell CM, Haythornthwaite JA, Edwards RR, Smith MT. Discordance between pain and radiographic severity in knee osteoarthritis: findings from quantitative sensory testing of central sensitization. Arthritis Rheum. 2013 Feb;65(2):363-72. doi: 10.1002/art.34646. PMID 22961435
- [Background] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Background] Imamura M, Imamura ST, Kaziyama HH, Targino RA, Hsing WT, de Souza LP, Cutait MM, Fregni F, Camanho GL. Impact of nervous system hyperalgesia on pain, disability, and quality of life in patients with knee osteoarthritis: a controlled analysis. Arthritis Rheum. 2008 Oct 15;59(10):1424-31. doi: 10.1002/art.24120. PMID 18821657
- [Background] Arendt-Nielsen L, Nie H, Laursen MB, Laursen BS, Madeleine P, Simonsen OH, Graven-Nielsen T. Sensitization in patients with painful knee osteoarthritis. Pain. 2010 Jun;149(3):573-581. doi: 10.1016/j.pain.2010.04.003. Epub 2010 Apr 24. PMID 20418016
- [Background] Gwilym SE, Oag HC, Tracey I, Carr AJ. Evidence that central sensitisation is present in patients with shoulder impingement syndrome and influences the outcome after surgery. J Bone Joint Surg Br. 2011 Apr;93(4):498-502. doi: 10.1302/0301-620X.93B4.25054. PMID 21464489
- [Background] Coombes BK, Bisset L, Vicenzino B. Cold hyperalgesia associated with poorer prognosis in lateral epicondylalgia: a 1-year prognostic study of physical and psychological factors. Clin J Pain. 2015 Jan;31(1):30-5. doi: 10.1097/AJP.0000000000000078. PMID 24480912
- [Background] Wylde V, Palmer S, Learmonth ID, Dieppe P. The association between pre-operative pain sensitisation and chronic pain after knee replacement: an exploratory study. Osteoarthritis Cartilage. 2013 Sep;21(9):1253-6. doi: 10.1016/j.joca.2013.05.008. PMID 23973138
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Peters TJ, Sanders C, Dieppe P, Donovan J. Factors associated with change in pain and disability over time: a community-based prospective observational study of hip and knee osteoarthritis. Br J Gen Pract. 2005 Mar;55(512):205-11. PMID 15808036
- [Background] Sterling M, Jull G, Vicenzino B, Kenardy J. Sensory hypersensitivity occurs soon after whiplash injury and is associated with poor recovery. Pain. 2003 Aug;104(3):509-517. doi: 10.1016/S0304-3959(03)00078-2. PMID 12927623
- [Background] Smart KM, Blake C, Staines A, Thacker M, Doody C. Mechanisms-based classifications of musculoskeletal pain: part 1 of 3: symptoms and signs of central sensitisation in patients with low back (+/- leg) pain. Man Ther. 2012 Aug;17(4):336-44. doi: 10.1016/j.math.2012.03.013. Epub 2012 Apr 23. PMID 22534654
- [Background] Yarnitsky D, Granot M, Granovsky Y. Pain modulation profile and pain therapy: between pro- and antinociception. Pain. 2014 Apr;155(4):663-665. doi: 10.1016/j.pain.2013.11.005. Epub 2013 Nov 21. No abstract available. PMID 24269491
- [Background] O'Neill S, Manniche C, Graven-Nielsen T, Arendt-Nielsen L. Association between a composite score of pain sensitivity and clinical parameters in low-back pain. Clin J Pain. 2014 Oct;30(10):831-8. doi: 10.1097/AJP.0000000000000042. PMID 24121529
- [Background] Wylde V, Palmer S, Learmonth ID, Dieppe P. Somatosensory abnormalities in knee OA. Rheumatology (Oxford). 2012 Mar;51(3):535-43. doi: 10.1093/rheumatology/ker343. Epub 2011 Nov 24. PMID 22120461
- [Background] Graven-Nielsen T, Wodehouse T, Langford RM, Arendt-Nielsen L, Kidd BL. Normalization of widespread hyperesthesia and facilitated spatial summation of deep-tissue pain in knee osteoarthritis patients after knee replacement. Arthritis Rheum. 2012 Sep;64(9):2907-16. doi: 10.1002/art.34466. PMID 22421811
- [Background] Cruz-Almeida Y, Fillingim RB. Can quantitative sensory testing move us closer to mechanism-based pain management? Pain Med. 2014 Jan;15(1):61-72. doi: 10.1111/pme.12230. Epub 2013 Sep 6. PMID 24010588
- [Background] Yunus MB. Central sensitivity syndromes: a new paradigm and group nosology for fibromyalgia and overlapping conditions, and the related issue of disease versus illness. Semin Arthritis Rheum. 2008 Jun;37(6):339-52. doi: 10.1016/j.semarthrit.2007.09.003. Epub 2008 Jan 14. PMID 18191990
- [Background] Staud R. Abnormal endogenous pain modulation is a shared characteristic of many chronic pain conditions. Expert Rev Neurother. 2012 May;12(5):577-85. doi: 10.1586/ern.12.41. PMID 22550986
- [Derived] O'Leary H, Smart KM, Moloney NA, Blake C, Doody CM. Pain sensitisation and the risk of poor outcome following physiotherapy for patients with moderate to severe knee osteoarthritis: protocol for a prospective cohort study. BMJ Open. 2015 Jun 9;5(6):e007430. doi: 10.1136/bmjopen-2014-007430. PMID 26059523